CLINICAL TRIAL: NCT01421966
Title: A Phase III Multicenter, Randomized, Double-Blind, Parallel-Group, Sham-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of CureXcell® as an Adjunct to Good Wound Care in Lower Extremity Chronic Ulcers in Adults With Diabetes Mellitus
Brief Title: Evaluation of CureXcell® in Treating Lower Extremity Chronic Ulcers in Adults With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Macrocure Ltd. (Industry)
Collaborators: Amarex Clinical Research (Other); ICON plc (Industry); ARANZ Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC-102
Record Dates: First submitted 2011-08-21; First posted 2011-08-23 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Lower Extremity Chronic Ulcers in Diabetics
Keywords: chronic ulcers; diabetic foot ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CureXcell® (Experimental)
  Interventions: Biological: CureXcell®
- Sham injection (Sham Comparator)
  Interventions: Biological: Sham injection

INTERVENTIONS:
Biological: CureXcell® — CureXcell® injection will be administered about every 4 weeks for up to 4 treatments, or until until ulcer closure, whichever occurs first.
  Arms: CureXcell®
Biological: Sham injection — The sham injections will be made by pressing on the ulcer with a needle connected to an empty syringe, at each cm of the ulcer bed
  Arms: Sham injection

SUMMARY:
Chronic foot ulcers are particularly prevalent in patients with underlying diabetes mellitus. These ulcers are reported to be the leading cause of hospitalization among people with diabetes.

The purpose of this study is to evaluate CureXcell® in treating chronic lower extremity ulcers in adults with diabetes mellitus. CureXcell® is a cell based therapy, containing activated homologous white blood cells prepared from donated healthy whole blood. A total of 280 patients will be randomized to receive either CureXcell® or sham.

DETAILED DESCRIPTION:
Chronic foot ulcers are particularly prevalent in patients with underlying diabetes mellitus. The prevalence of diabetes mellitus is growing at epidemic rates in Europe, United States and in general worldwide. Foot ulceration is a serious complication of diabetes mellitus associated with increased risk of infection, gangrene and amputation. These ulcers are reported to be the leading cause of hospitalization among people with diabetes. Despite existing ulcer therapies and technologies, there continues to be a great necessity for new wound healing technologies that will further improve healing rates for these chronic ulcers that remain a major source of morbidity, concern, and cost. This Phase 3 multinational, multicenter, randomized, double-blind, controlled study is designed to evaluate CureXcell® in treating lower extremity chronic ulcers in adults with Diabetes Mellitus.

CureXcell® is a cell based therapy obtained from donated whole blood. The blood are collected from healthy, young adult (age 18-40), the cells separated and then activated by hypo-osmotic shock.

A total of 280 patients, in approximately 35 sites in the US, Canada and Israel, will be randomized to receive either CureXcell® or control.

The primary objective of the study is to evaluate the clinical benefit of CureXcell® (study biologic) compared to control, as adjunct to Good Ulcer Care. Additional objectives are to demonstrate safety, tolerability and durability of CureXcell® compared to control.

The study has two phases: a core double-blind phase and a follow up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years of age with diabetes type 1 or type 2;
2. Patients with HbA1c ≤ 12%;
3. Patients with at least one lower extremity (on or below the malleolus (ankle bone)), at least full-thickness ulcer (penetrating through the whole layer of the skin), which has been unresponsive to any treatment for at least 4 weeks;
4. Ulcers with an area between ≥ 1 cm2 and ≤ 20 cm2 (after sharp debridement of free, non-viable, hyperkeratotic and fibrotic tissue to the extent possible);
5. Ankle Brachial Index ≥ 0.65;

Exclusion Criteria:

1. Patients with more than two ulcers on the same foot or more than a total of three chronic ulcers;
2. Patients with ulcers primarily caused by venous insufficiency;
3. Patients whose target ulcer has decreased > 25% in size from screening to baseline;
4. Malignancy within the past 5 years excluding successfully treated basal cell carcinoma;
5. Significantly compromised immunity for any reason including radiation therapy, chemotherapy or HIV;
6. Current clinical osteomyelitis;
7. Acute Charcot foot;
8. Current sepsis;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete healing/closure of their target ulcer at any time during the 16-week double-blind core treatment period with sustained complete closure for 4 additional weeks of follow-up. | up to 20 weeks

SECONDARY OUTCOMES:
Time to complete closure of the Target Ulcer during the core double blind treatment phase with sustained complete closure for 4 additional weeks of follow-up. | up to 20 weeks
Proportion of patients with at least 50% closure of target ulcer during the 16-week core treatment period. | 16 weeks
Proportion of patients whose Target Ulcer completely closed during the core double blind treatment phase and remained closed at the FU12 follow-up visit. | up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vickie Driver, MS, DPM, FACFAS, Principal Investigator — VA New England Health Care Division
Locations (37):
- United States (31):
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fresno, California
  - San Francisco, California
  - Sylmar, California
  - Gulf Breeze, Florida
  - Hialeah, Florida
  - Miami, Florida
  - South Miami, Florida
  - Evans, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Oak Park, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Toms River, New Jersey
  - Mineola, New York
  - New York, New York
  - Lima, Ohio
  - Aiken, South Carolina
  - Greenville, South Carolina
  - Dallas, Texas
  - Lewisville, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
- Canada (2):
  - Winnipeg, Manitoba
  - Boucherville, Quebec
- Israel (4):
  - Haifa
  - Holon
  - Jerusalem
  - Tel Aviv